CLINICAL TRIAL: NCT06528691
Title: PHASE 2 Study of Entrectinib as a Single Agent in Upfront Therapy for Children <3 Years of Age With NTRK1/2/3 or ROS1-FUSED CNS Tumors (GLOBOTRK)
Brief Title: Entrectinib as a Single Agent in Upfront Therapy for Children <3 Years of Age With NTRK1/2/3 or ROS1-FUSED CNS Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLOBOTRK; NCI-2024-02977 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-07-22; First posted 2024-07-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: High Grade Glioma; CNS Tumor
Keywords: CNS Tumors; High Grade Glioma with NTRK1/2/3 gene fusion; High Grade Glioma with ROS1 gene fusion; CNS tumor other than HGG harboring NTRK1/2/3 gene fusion; CNS tumor other than HGG harboring ROS1 gene fusion; Children
MeSH Terms: conditions — Glioma; Central Nervous System Neoplasms | interventions — entrectinib; Cyclophosphamide; Etoposide; Carboplatin; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Pediatric patients <3 years of age, with NTRK1/2/3 or ROS1-fused high-grade gliomas and other CNS tumors will be treated with frontline single-agent entrectinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entrectinib therapy, Cohort 1 and Cohort 2 (Experimental): Cohort 1: Patients who are younger than 3 years of age diagnosed with NTRK1/2/3- or ROS1-fused high-grade glioma (HGG) will receive therapy as outline in Detailed Description.
  Cohort 2: Patients who are younger than 3 years of age diagnosed with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG will receive therapy as outline in Detailed Description.
  Interventions: Drug: Entrectinib; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Carboplatin; Biological: G-CSF; Biological: Pegfilgrastim; Procedure: Surgery

INTERVENTIONS:
Drug: Entrectinib — Given orally (PO) or enterally
  Other Names: Rozlytrek
Drug: Cyclophosphamide — Given intravenous (IV)
  Other Names: Cytoxan®
Drug: Etoposide — Given IV
  Other Names: VP-16
Drug: Carboplatin — Given IV
  Other Names: Paraplatin®
Biological: G-CSF — Given subcutaneous (SQ) or IV
  Other Names: Filgrastim
Biological: Pegfilgrastim — Given SQ as part of recommended Bridging Therapy instead of G-CSF.
  Other Names: Neulasta
Procedure: Surgery — A gross total resection or significant debulking may become possible if a response to entrectinib is seen.
  Other Names: Surgical resection

SUMMARY:
This clinical trial tests how well entrectinib works to treat patients less than 3 years of age with NTRK 1/2/3 or ROS1 fused, high grade glioma or other central nervous system (CNS) tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

* To determine the overall response rate of entrectinib when used as first line therapy in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused high-grade glioma (HGG) (Cohort 1).

SECONDARY OBJECTIVES

* To estimate the 2-year and 5-year progression free survival (PFS) and overall survival (OS) in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused HGG treated with entrectinib as first line therapy (Cohort 1).
* To estimate the duration of response (DOR) in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused HGG treated with entrectinib as first line therapy (Cohort 1).
* To evaluate the fraction of patients with NTRK1/2/3- or ROS1-fused HGG treated who have second surgeries and a gross-total resection after treatment with entrectinib is achieved, overall and by country and hospital (Cohort 1).
* To describe the overall response rate of entrectinib when used as first line therapy in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG (Cohort 2).
* To estimate the 2-year and 5-year PFS and OS in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG treated with entrectinib as first line therapy (Cohort 2).
* To estimate the duration of response (DOR) in patients who are younger than 3 years of age with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG treated with entrectinib as first line therapy (Cohort 2).
* To evaluate the fraction of patients with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG who have second surgeries and a gross-total resection after treatment with entrectinib is achieved, overall and by country and hospital (Cohort 2).
* To describe toxicities experienced by patients younger than 3 years of age treated with entrectinib (Cohort 1 and 2).
* To evaluate number of patients that are screened for the study and eligible versus enrolled and treated with entrectinib (Cohort 1 and 2).
* To measure the time intervals (days) from time of initial diagnostic surgery to screening and enrollment in this study (Cohort 1 and 2).

The trial will have 2 cohorts: Cohort 1: patients diagnosed with NTRK1/2/3- or ROS1-fused high-grade glioma (HGG) and Cohort 2: patients diagnosed with NTRK1/2/3- or ROS1-fused CNS tumors other than HGG.

Patients receive entrectinib enterally once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients requiring bridging therapy prior to starting entrectinib may receive cyclophosphamide intravenously (IV) over 1 hour on day 1, etoposide IV over 1 hour on day 1 and 2, carboplatin IV over 1 hour on day 2, filgrastim subcutaneously (SC) or IV or pegfilgrastim SC on day 3.

A gross total resection or significant debulking may become possible if a response to entrectinib is seen. If surgical resection is performed and a gross total resection is achieved, 24 cycles of entrectinib will be completed, including those before and after surgery.

After treatment, patients will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria: Screening Phase

* Age from birth to age <3 years at the time of diagnosis (date of surgical resection/biopsy)
* Participant with presumed newly diagnosed tumor in the supratentorial compartment
* Patient must have measurable disease based on RAPNO criteria
* ≤84 days since surgery (resection or biopsy)
* Available tumor tissue for central review
* Parent/guardian has the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines

Exclusion Criteria: Screening Phase

* Previous exposure to cytotoxic chemotherapy or radiotherapy

Inclusion Criteria: COHORT 1

* Patients must be <3 years of age at the time of diagnosis (date of surgical resection/biopsy)
* High-grade glioma (World Health Organization [WHO] grade III or IV) harboring NTRK1/2/3 or ROS1 gene fusions as determined by central pathology review
* Patients must have measurable disease as defined by RAPNO criteria
* Patients are eligible at the time of diagnosis, prior to any exposure to chemotherapy, targeted therapy, immunotherapy, cellular therapy or radiation
* ≤28 days since study screening
* Lansky score ≥50% and a minimum life expectancy of ≥ 12 weeks
* Neurologic deficits must have been stable for at least 7 days prior to study enrollment
* Hemoglobin ≥ 8 g/dL (without transfusion or erythropoietin use within 7 days prior to enrollment)
* Platelet count ≥ 75,000/µL (without transfusion within 7-day period prior to enrollment)
* Absolute neutrophil count >1,000/µL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x the upper limit of normal (ULN)
* Bilirubin ≤ 1.5 x ULN
* Adequate renal function as defined by the following age-based serum creatinine concentrations:

  * 0 to <1 year: 0.5 mg/dL
  * 1 to <2 years: 0.6 mg/dL
  * 2 to 3 years: 0.8 mg/dL
* Adequate cardiac function as defined by electrocardiogram (ECG) with Fridericia's corrected QT interval (QTc) ≤ 450 msec and echocardiogram left ventricular ejection fraction (LVEF) >50%
* Screening and enrollment consents signed
* Willingness and ability to comply with treatment plan, scheduled visits, laboratory tests and other study procedures

Inclusion Criteria: COHORT 2

* Patients must be <3 years of age at the time of diagnosis (date of surgical resection/biopsy)
* CNS tumor other than HGG harboring NTRK1/2/3 or ROS1 gene fusions as determined by central pathology review
* Patients must have measurable disease as defined by RAPNO criteria
* Patients are eligible at the time of diagnosis, prior to any exposure to chemotherapy, targeted therapy, immunotherapy, cellular therapy or radiation
* ≤28 days since study screening
* Lansky score ≥50% and a minimum life expectancy of ≥ 12 weeks
* Neurologic deficits must have been stable for at least 7 days prior to study enrollment.
* Hemoglobin ≥ 8 g/dL (without transfusion or erythropoietin use within 7 days prior to enrollment)
* Platelet count ≥ 75,000/µL (without transfusion within 7-day period prior to enrollment);
* Absolute neutrophil count >1,000/µL.
* ALT and ALT ≤2.5x the upper limit of normal (ULN)
* Bilirubin ≤ 1.5 x ULN
* Adequate renal function as defined by the following age-based serum creatinine concentrations:

  * 0 to <1 year: 0.5 mg/dL
  * 1 to <2 years: 0.6 mg/dL
  * 2 to 3 years: 0.8 mg/dL
* Adequate cardiac function as defined by ECG with QTc ≤ 450 msec and echocardiogram LVEF >50%
* Screening and enrollment consents signed
* Willingness and ability to comply with treatment plan, scheduled visits, laboratory tests and other study procedures

Exclusion Criteria: COHORT 1 AND 2

* Clinically significant medical disorder that could compromise the ability to tolerate study therapy or would interfere with the study procedures or results history
* History of recent (3 months) symptomatic congestive heart failure
* Known active, uncontrolled infection (bacterial, fungal, or viral)
* Receiving enzyme inducing antiepileptic drugs (EIAEDs)
* Any prior cancer therapy including chemotherapy (excluding Bridging Chemotherapy Cycle), targeted therapy, immunotherapy, cellular therapy, or radiation
* Receiving another investigational agent concurrently
* Surgery within 2 weeks prior to treatment enrollment
* Patients with known hypersensitivity to excipients of the investigational medicinal product
* Active gastrointestinal disease or malabsorption disorder (e.g. Crohn's disease, ulcerative colitis, short-gut syndrome) that would impair drug absorption
* Inability to take medication enterally

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Cohort 1) | After cycle 4 (each cycle is 28 days).
  ORR is defined as the percentage of patients with either partial or complete response assessed at the protocol-defined evaluation timepoint. Overall response will be determined by the central imaging review based on the scheduled evaluations.

SECONDARY OUTCOMES:
Progression free survival (PFS) (Cohort 1) | At 2 and 5 years
  PFS is defined as the time from initiation of protocol treatment to first event (progressive disease, death due to any cause), or date last follow-up among those who have not had an event. Described using Kaplan Meier method.
Overall survival (OS) (Cohort 1) | At 2 and 5 years
  OS is defined as the time from date of diagnosis to date of death due to any cause or date last follow-up. Described using Kaplan Meier method.
Duration of response (DOR) (Cohort 1) | Up to 5 years
  DOR is defined as time from date of first response (partial or complete) until the date of progression or last follow-up. Described as median time.
Patients who have second surgeries (Cohort 1) | Up to 5 years
  Percentage of patients who had second surgeries.
Patients who undergo gross-total resection after treatment (Cohort 1) | Up to 5 years
  Percentage of patients who underwent a gross-total resection.
ORR (Cohort 2) | After cycle 4 (each cycle is 28 days).
  ORR is defined as the percentage of patients with either partial or complete response assessed at the protocol-defined evaluation timepoint. Overall response will be determined by the central imaging review based on the scheduled evaluations.
PFS (Cohort 2) | At 2 and 5 years
  PFS is defined as the time from initiation of protocol treatment to first event (progressive disease, death due to any cause), or date last follow-up among those who have not had an event. Described using Kaplan Meier method.
OS (Cohort 2) | At 2 and 5 years
  OS is defined as the time from date of diagnosis to date of death due to any cause or date last follow-up. Described using Kaplan Meier method.
DOR (Cohort 2) | Up to 5 years
  DOR is defined as time from date of first response (partial or complete) until the date of progression or last follow-up. Described as median time.
Patients who have second surgeries (Cohort 2) | Up to 5 years
  Percentage of patients who had second surgeries. [Time Frame: Up to 5 years]
Patients who undergo gross-total resection after treatment (Cohort 2) | Up to 5 years
  Percentage of patients who underwent a gross-total resection.
Incidence of adverse events (Cohort 1 and 2) | Up to 5 years
  Percentage of adverse events on therapy including Entrectinib, captured using National Cancer Institute Common Terminology Criteria for Adverse Events 5.0.
Number of patients screened versus enrolled and treated (Cohort 1 and 2) | Up to 5 years
  Number of enrolled and treated patients as a percentage of number of patients screened and eligible for study.
Time from initial diagnostic surgery to screening and enrollment (Cohort 1 and 2) | Up to 5 years
  Median time in days from initial surgery to screening and enrollment on study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moreira, MD, MEd, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols